CLINICAL TRIAL: NCT04163029
Title: Analysis of the Impact on the Incidence of Postoperative Infections (at the Surgical Site, Flap and Lung) and on the Length of Stay of Oral Care Before Surgery on the ENT Sphere With Flap Reconstruction
Brief Title: Oral Care Study of Postoperative Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Other Study IDs: RAACBPTM
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cancer, Mouth
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- preoperative oral care
  Interventions: Procedure: Preoperative oral care

INTERVENTIONS:
Procedure: Preoperative oral care — tooth brushing and mouthwash with chlorhexidine 0,2% five day before surgery

SUMMARY:
Reduce the incidence of post-operative infections after ENT surgery and flap reconstruction by performing preoperative oral and dental care

DETAILED DESCRIPTION:
Reduce the incidence of post-operative infections after ENT surgery and flap reconstruction by performing preoperative oral and dental care

ELIGIBILITY:
Inclusion Criteria:

* ENT surgery with free flap reconstruction

Exclusion Criteria:

* Allergy to chlorhexidine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients operated on for transmandibulary buccopharyngectomy with recognition, free flap struction
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-22 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative infections | through study completion, an average of 1 year
  incidence of postoperative infections

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Javillier, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- University of Liege, University Hospital, Liège, Belgium